CLINICAL TRIAL: NCT04169724
Title: Feasibility of The Mindfulness Meditation App "Calm" to Reduce Burnout in Physician Assistant Students
Brief Title: Meditation for Burnout in PA Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: Calm.com, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00010572
Record Dates: First submitted 2019-11-18; First posted 2019-11-20 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Burnout, Student; Feasibility
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Calm (Experimental): Participants will be asked to download the Calm app on their smartphone. Participants will then receive an email containing login credentials to access the Calm app. Once they receive this email and they receive their study start date, they will be asked to meditate for at least 10 minutes a day for 8 weeks. This prescription mimics how a new, paying member would use the app. Participants in the intervention group will be emailed weekly reminders.
  Interventions: Behavioral: Calm Meditation
- Waitlist (No Intervention): Participants randomized to the control group will be asked to maintain their normal routine for 8 weeks and to avoid using the Calm meditation app.

INTERVENTIONS:
Behavioral: Calm Meditation — 10 minutes per day of meditation via the Calm app.
  Arms: Calm

SUMMARY:
This study investigates the feasibility and effects of an app-based mindfulness meditation intervention for PA students.

DETAILED DESCRIPTION:
The purpose of this study is to determine the feasibility of an app-based mindfulness meditation intervention for PA students.

The investigators will measure feasibility of using the Calm app for 10-minutes a day for four weeks in PA students. Feasibility will be measured with acceptability (i.e. satisfaction survey), demand (participation in the app as prescribed), and practicality (i.e., survey). Secondly, the investigators will determine the preliminary effects of a 4-week meditation intervention on burnout levels in PA students when compared to a wait list control group. Burnout symptoms (primary outcome), mindfulness, stress levels, and depressive symptoms (secondary outcomes) will be measured at baseline and post-intervention (4-weeks). Data gathered from this study will inform a future randomized controlled trial to determine the effects of a mindfulness meditation app on burnout in PA students. The information could also be used to design other studies assessing burnout in the workplace.

Aim 1: Determine the feasibility (acceptability, demand, practicality) of using the Calm app 10-minutes per day for four weeks in PA students. For the intervention group, our benchmarks will be as follows: 1) Acceptability (i.e., satisfaction) ≥70%, 2) Demand (i.e., participation in the app as prescribed, intention to use) ≥70%, 3) Practicality (i.e., survey) ≥70%.

Aim 2: Determine the preliminary effects of using the Calm app 10-minutes per day for four weeks on burnout (primary outcome) mindfulness, stress levels, and depressive symptoms (secondary outcomes) in PA students as compared to a wait-list control group.

ELIGIBILITY:
Inclusion Criteria:

* Physician assistant students currently enrolled in school who do not practice meditation regularly
* > 18 years of age
* Able to speak/read/understand English
* Residing in the U.S.
* Regular internet access via mobile phone, tablet, etc.
* Willing to participate in app-based meditation program
* Burnout, classified as a score greater than or equal to 3 on the non-propriety single item burnout measure.

Exclusion Criteria:

* Physician assistant students who currently (within the last six months) practice meditation
* Professionals who identify as a practicing physician assistant
* People who are not currently enrolled in physician assistant school
* Individuals who are not burnt out, classified as a score less than or equal to 2 on the non-propriety single item burnout measure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2020-03-09 (Actual); Study Completion 2020-03-09 (Actual)

PRIMARY OUTCOMES:
Burnout | Change from baseline to post-intervention (week 4).
  The Maslach Burnout Inventory is a 22-item inventory used to measure aspects of the burnout syndrome within three subscales: emotional exhaustion, depersonalization, and personal accomplishment. Using a seven-point scale (0, never; 1, a few times per year; 2, once a month; 3, a few times a month; 4, once a week; 5, a few times a week; 6, every day), participants rate their experience of burnout. Possible scores on the emotional exhaustion subscale range from 0 to 54. Possible scores on the depersonalization subscale range from 0 to 30. For both the emotional exhaustion and depersonalization subscales, higher mean scores correspond to higher degrees of burnout. Possible scores on the personal accomplishment subscale range from 0 to 48. Lower mean scores on the personal accomplishment subscale correspond to higher degrees of burnout. Scores are computes via sum.

SECONDARY OUTCOMES:
Mindfulness | Change from baseline to post-intervention (week 4).
  The Freidburg Mindfulness Inventory is used to measure mindfulness using a 14-item questionnaire covering all aspects of mindfulness. Using a four-point scale, (1, rarely; 2, occasionally; 3, fairly often; 4, almost always), participants are asked to characterize their experience of mindfulness. Higher scores indicate higher levels of mindfulness. Scores are computed via sum.
Stress | Change from baseline to post-intervention (week 4).
  The Perceived Stress Scale is a 10-item inventory used for the assessment of perceived stress. The scale measures the degree to which situations are appraised as stressful. The items are rated on a 5-point Likert scale ranging from 0 (never) to 4 (very often). Higher scores indicate higher levels of stress. Scores are computed via sum.
Depression | Change from baseline to post-intervention (week 4).
  The Patient Health Questionnaire-9 is used to measure and diagnose depression using a 9-item self-report measure. Items are rated 4-item scale ranging from 0 (Not at all) to 3 (nearly every day). Higher scores correspond with more severe depressive symptoms. Scores are computed via sum.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Huberty, PhD, Principal Investigator — Arizona State University
Locations (1):
- Arizona Biomedical Collaborative, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No